CLINICAL TRIAL: NCT05843955
Title: Assessment of Non-alcoholic Fatty Liver Disease and Risk Factors in Women With Polycystic Ovary Syndrome
Brief Title: Non-alcoholic Fatty Liver Disease in Women With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Principal Investigator, Hacettepe University
Other Study IDs: GO 15/547
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: PCOS; NAFLD
Keywords: polycystic ovary syndrome; non-alcoholic fatty liver disease; obesity; insulin resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Polycystic Ovary Syndrome; Obesity; Insulin Resistance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Polycystic ovary syndrome (PCOS): PCOS was diagnosed according to the revised 2003 Rotterdam Consensus as the presence of at least two of the following three criteria: (i)oligomenorrhoea or anovulation; (ii)clinical and/or biochemical signs of hyperandrogenemia and (iii)polycystic ovaries on ultrasound.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Nutritional status, physical activity levels, anthropometric measurements, and biochemical parameters of individuals were examined. A food consumption frequency questionnaire was administered.

SUMMARY:
This study was planned to examine the prevalence of vitamin D insufficiency, insulin resistance, non-alcoholic fatty liver disease (NAFLD), and their relationship with each other and the nutritional status of individuals with polycystic ovary syndrome (PCOS) in reproductive age, by evaluating anthropometric, biochemical, and ultrasonographic findings and food consumption frequency data.

DETAILED DESCRIPTION:
A total of 72 female individuals diagnosed with PCOS were included in the study. Nutritional status, physical activity levels, anthropometric measurements, and biochemical parameters of individuals were examined. A food consumption frequency questionnaire was applied to the individuals. According to the 2003 Rotterdam Consensus revision, PCOS is diagnosed when at least two of the following three conditions are present: Polycystic ovaries on ultrasonography, oligomenorrhoea, or anovulation; clinical and/or biochemical symptoms of hyperandrogenemia. Testing was done on insulin, lipid profiles, fasting plasma glucose, and liver function. Bioelectrical impedance analysis was used to determine body weight and composition. An abdominal ultrasound was used to diagnose NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* PCOS diagnosis
* no use of oral contraceptives or any hormone therapy in the last 3 months
* no use of vitamin D supplements in the last 3 months
* no use of oral antidiabetic drugs in the last 3 months

Exclusion Criteria:

* adrenal dysfunction
* diabetes mellitus
* pregnancy
* alcohol consumption
* a history of chronic viral hepatitis
* autoimmune liver disease
* other liver diseases
* history of hepatotoxicity
* use of antihypertensive, antidiabetic, lipid-lowering drugs

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The appropriate sample size was determined to be 65 using power analysis in accordance with the results of the prior studies, with a 90% confidence interval and a 0.05 type-I error. The Rotterdam Consensus, revised in 2003, defined polycystic ovary syndrome (PCOS) as the presence of at least two of the following three criteria: (i) oligomenorrhoea or anovulation; (ii) clinical and/or biochemical signs of hyperandrogenemia; and (iii) ultrasound-confirmed polycystic ovaries. 328 volunteer women who visited the clinic throughout the research period were chosen as participants after being screened for eligibility. This study included 72 women who were confirmed to be eligible and ranged in age from 18 to 40.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D levels | 3 months
  Serum vitamin D levels were measured by immunoassay analyzer.
Insulin resistance | 3 months
  Insulin resistance analyzed by homeostasis model assessment-insulin resistance (HOMA-IR) formulation.
Non-alcoholic fatty liver disease (NAFLD) grade | 3 months
  NAFLD grade was evaluated by ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Nutrition and Dietetics Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to ethical concerns.